CLINICAL TRIAL: NCT02962661
Title: Randomized 3-Arm Trial With Standard of Care Alone vs Either Intravenous Infusion or Transendocardial Injection of Allogeneic Bone Marrow Derived Multipotent Mesenchymal Stromal Cells (MSCs) Plus Standard of Care in Patients With Anthracycline-Associated Cardiomyopathy
Brief Title: Donor Bone Marrow Derived Mesenchymal Stem Cells in Controlling Heart Failure in Patients With Cardiomyopathy Caused by Anthracyclines
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0835; NCI-2016-01921 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0835 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cardiomyopathy; Heart Failure; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (hMSCs IV) (Experimental): Patients receive hMSCs IV over 10-20 minutes on days 1, 14, 21, and 28 and standard of care treatment for heart failure in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Best Practice; Other: Laboratory Biomarker Analysis; Drug: Mesenchymal Stem Cell Transplantation
- Arm II (hMSCs transendocardially) (Experimental): Patients receive hMSCs transendocardially for a total of 15 injections and standard of care treatment for heart failure in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Best Practice; Other: Laboratory Biomarker Analysis; Drug: Mesenchymal Stem Cell Transplantation
- Arm III (standard of care) (Active Comparator): Patients receive standard of care treatment for heart failure.
  Interventions: Other: Best Practice; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Best Practice — Given standard of care
  Other Names: standard of care; standard therapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mesenchymal Stem Cell Transplantation — Given IV
  Arms: Arm I (hMSCs IV)
Drug: Mesenchymal Stem Cell Transplantation — Given transendocardially
  Arms: Arm II (hMSCs transendocardially)

SUMMARY:
This randomized pilot phase I trial studies the side effects of donor bone marrow derived mesenchymal stem cells in controlling heart failure in patients with cardiomyopathy caused by anthracyclines. Donor bone marrow derived mesenchymal stem cells may help to control symptoms of heart failure and improve heart function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate the safety of allogeneic human mesenchymal stem cells (hMSCs) administered by intravenous infusion and transendocardial injection in patients with left ventricular (LV) dysfunction and heart failure secondary to chemotherapy with anthracyclines.

SECONDARY OBJECTIVE:

I. To demonstrate the efficacy of allogeneic hMSCs administered by intravenous infusion and transendocardial injection in patients with left ventricular dysfunction (left ventricular ejection fraction [LVEF] < 40%) and heart failure secondary to treatment with anthracyclines.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive hMSCs intravenously (IV) over 10-20 minutes on days 1, 14, 21, and 28 and standard of care treatment for heart failure in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive hMSCs transendocardially for a total of 15 injections and standard of care treatment for heart failure in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive standard of care treatment for heart failure.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with LVEF </= 40% documented from treatment with anthracyclines for any malignancy at any dose at any time without evidence of other causes of cardiomyopathy.
2. Age >/= 18 and </= 90 years of age. English and non-English speaking patients are eligible.
3. Documented NYHA class I, II and III.
4. For patients who have received trastuzumab: Persistent LV dysfunction must be present 90 days after discontinuation of trastuzumab.
5. Able to perform 6 minute walk test.
6. Been treated with appropriate maximal medical therapy for heart failure.
7. Patient or legally authorized representative able to sign informed consent.

Exclusion Criteria:

1. Evidence of Ischemic Heart Disease as determined by study cardiologist.
2. Significant Valvular Disease. (AS with AVA <1.5 and severe AR and MR)
3. History of Familial Cardiomyopathy.
4. Recent documented myocarditis within 2 months of enrollment.
5. History of Infiltrative cardiomyopathy or restrictive cardiomyopathy.
6. Presence of left ventricular thrombus as documented by echocardiography or left ventriculogram.
7. Liver function tests > 3 x upper limit of normal.
8. NYHA class IV heart failure.
9. Inotropic dependence.
10. Unstable or life-threatening arrhythmia.
11. For patients not on anticoagulants, INR>1.5
12. Mechanical or Bioprosthetic heart valve.
13. Cardiogenic shock.
14. Breastfeeding and/or pregnant women.
15. Autoimmune disorders on current immunosuppressive therapy.
16. Active infection not responding to appropriate therapy as determined by Study Chair.
17. Trastuzumab treatment within the last 3 months.
18. Automatic implantable cardioverter defibrillator (AICD) placement within the last 30 days.
19. AICD firing within the last 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-07-18 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Statistical analyses of safety will be descriptive.
Change in left ventricular ejection fraction (LVEF) | Baseline to 6 months
  The comparison will be between the two groups of patients.

SECONDARY OUTCOMES:
Change in improvement of left ventricular (LV) systolic function as assessed by LVEF | Baseline up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between each investigational group and the control group. If both investigation groups are significant at the p < .05 level, then the two investigational drugs can be compared using a gatekeeping procedure. These intervals and the associated p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
LV end-systolic and end-diastolic volumes as determined by contrast-enhanced 2-dimensional(D)/3D echography | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between each investigational group and the control group. If both investigation groups are significant at the p < .05 level, then the two investigational drugs can be compared using a gatekeeping procedure. These intervals and the associated p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Cardiac death | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between each investigational group and the control group. If both investigation groups are significant at the p < .05 level, then the two investigational drugs can be compared using a gatekeeping procedure. These intervals and the associated p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Re-hospitalization after heart failure | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between each investigational group and the control group. If both investigation groups are significant at the p < .05 level, then the two investigational drugs can be compared using a gatekeeping procedure. These intervals and the associated p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Aborted death from an automatic implantable cardioverter defibrillator (AICD) firing | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between each investigational group and the control group. If both investigation groups are significant at the p < .05 level, then the two investigational drugs can be compared using a gatekeeping procedure. These intervals and the associated p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Nonfatal myocardial infarction | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between each investigational group and the control group. If both investigation groups are significant at the p < .05 level, then the two investigational drugs can be compared using a gatekeeping procedure. These intervals and the associated p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.
Revascularization | Up to 6 months
  As regards statistical analyses, the results of the trial will be displayed in table format. Will provide confidence intervals of the differences in change from baseline between each investigational group and the control group. If both investigation groups are significant at the p < .05 level, then the two investigational drugs can be compared using a gatekeeping procedure. These intervals and the associated p-values will be calculated using two-sample t-tests, with no adjustments for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Olson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org